CLINICAL TRIAL: NCT07113301
Title: Evaluation of Agreement in Histological Findings Between Core Needle and Incisional Biopsies
Brief Title: Incisional Biopsy Versus Core-needle Biopsy in Bone Tumors Analysis
Acronym: INSPECTOR
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: INSPECTOR
Record Dates: First submitted 2025-07-30; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Malignant Bone Tumor
MeSH Terms: conditions — Bone Neoplasms | interventions — Biopsy, Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: incisional or core-needle biopsy for tumor diagnosis — incisional or core-needle biopsy for tumor diagnosis

SUMMARY:
The investigators will collect data of patients with high suspicion of malignant bone tumor based on radiological imaging who underwent/will undergo both core needle biopsy and incisional biopsy for diagnostic confirmation by histological examination.

From 01/01/2015 to the approval date of this study: retrospective study; from the approval date of this study to 31/12/2027: prospective study. the investigators expect to collect data from a total of 72 patients: approximately 30 patients for the retrospective study and 42 for the prospective study. A review will be made from the medical records, radiological imaging, and histological data of partecipants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years
* Patients with high suspicion of malignant bone tumor who underwent/will undergo both core needle biopsy and incisional biopsy
* Male and female patients treated at Rizzoli Orthopaedic Institute from the approval date of this study to 31/12/2027
* Patients with available clinical and imaging data

Exclusion Criteria:

* Patients with bone tumor who underwent/will undergo only core needle biopsy
* Patients with bone tumor who underwent/ will undergo only incisional biopsy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients surgically treated at Rizzoli Orthopaedic Institute from the approval date of this study to 31/12/2027
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
compare the agreement between core needle biopsy and incisional biopsy, based on Cohen's kappa coefficient. | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kasraeian S, Allison DC, Ahlmann ER, Fedenko AN, Menendez LR. A comparison of fine-needle aspiration, core biopsy, and surgical biopsy in the diagnosis of extremity soft tissue masses. Clin Orthop Relat Res. 2010 Nov;468(11):2992-3002. doi: 10.1007/s11999-010-1401-x. PMID 20512437
- [Background] Mitsuyoshi G, Naito N, Kawai A, Kunisada T, Yoshida A, Yanai H, Dendo S, Yoshino T, Kanazawa S, Ozaki T. Accurate diagnosis of musculoskeletal lesions by core needle biopsy. J Surg Oncol. 2006 Jul 1;94(1):21-7. doi: 10.1002/jso.20504. PMID 16788939
- [Background] Errani C, Traina F, Perna F, Calamelli C, Faldini C. Current concepts in the biopsy of musculoskeletal tumors. ScientificWorldJournal. 2013 Jun 5;2013:538152. doi: 10.1155/2013/538152. Print 2013. PMID 23844403